CLINICAL TRIAL: NCT05022121
Title: Integrated Supported Biopsychosocial Self-Management for Back Related Leg Pain
Acronym: SUPPORT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: University of Pittsburgh (Other); Duke University (Other); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CSH-2021-30117; R34AT011209 (NIH)
Record Dates: First submitted 2021-05-18; First posted 2021-08-26 (Actual); Results first posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-02

CONDITIONS: Low Back Pain; Sciatica; Back Related Leg Pain; Pain, Chronic; Intervertebral Disc Displacement
MeSH Terms: conditions — Low Back Pain; Sciatica; Chronic Pain; Intervertebral Disc Displacement

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supported Biopsychosocial Self-Management (SBSM) (Experimental): Supported Biopsychosocial Self-Management (SBSM)
  Interventions: Behavioral: Supported Biopsychosocial Self-Management (SBSM)
- Medical Care (Active Comparator): Medical Care
  Interventions: Drug: Medical Care

INTERVENTIONS:
Behavioral: Supported Biopsychosocial Self-Management (SBSM) — Participants receive training and instruction in skills to engage in healthy physical, psychological, and social self-management behaviors. This will be accomplished through 6-12 sessions with a trained chiropractor or physical therapist. Patients will receive training and instruction in exercises targeting posture, strength, stabilization, and mobility based on their individual needs. They will learn psychological strategies including problem solving and cognitive restructuring to address unhelpful thoughts and emotions. Social strategies include pleasant activity planning with a social focus, and communication techniques for navigating relationships to garner support for self-sufficiency. Other elements include providing key evidence based information about BRLP and spinal manipulation therapies (SMT). SMT will include manipulation, mobilization and soft-tissue treatment. Other intervention elements include enablement, persuasion, and resources and materials to support the patient.
  Arms: Supported Biopsychosocial Self-Management (SBSM)
Drug: Medical Care — Medical care will be comprised of primarily medication management, which is a standard first-line approach for back-related leg pain in primary care. Choice of medications is informed by the current evidence and the American College of Physicians guidelines on noninvasive treatment for LBP which balances evidence for risks and benefits when making recommendations. Decisions regarding medication selection will be made collaboratively between the study provider and patient after a discussion of risk/benefit profiles and patient preferences, including prior response. Study providers licensed to prescribe FDA-approved medications will call-in the prescription for the medication of choice to the participant's preferred pharmacy, as is typical in clinical practice.
  Arms: Medical Care

SUMMARY:
Guidelines advocate several complementary modalities as alternatives to drugs and other invasive treatments for chronic low back pain (LBP) conditions. However, there is little high-quality research investigating treatments for back-related leg pain, one of the more severe and disabling presentations of LBP. The investigators are conducting a pilot study to assess the feasibility of a future phase II multi-site randomized clinical trial (RCT). The future trial will assess the comparative effectiveness of a novel supported biopsychosocial self-management (SBSM) intervention versus Medical Care (MC).

ELIGIBILITY:
Inclusion Criteria:

* Back-related leg pain (BRLP) consistent with the Quebec Task Force (QTF) classifications 2-4 (radiating pain into proximal or distal extremity with or without neurological signs).
* 18 years of age or older.
* Back-related leg pain severity of 3 or higher at all screening assessments (0 to 10 scale)
* Episode duration of 12 weeks or more
* Ability to read English fluently

Exclusion Criteria:

* Spinal stenosis (QTF 7)
* Specific, non-mechanical causes of BRLP (QTF 11; e.g. infection, tumor)
* Contraindications to study interventions (e.g. spinal fracture (QTF 5))
* Inflammatory conditions of the lumbar spine (QTF 11)
* Lumbar fusion
* Progressive neurological deficits
* Cauda equina syndrome
* Pregnancy, nursing
* Ongoing care from another healthcare provider for BRLP
* Severe unmanaged comorbid conditions (e.g. substance abuse, major depressive disorder, stage 3 hypertension).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2022-01-26 (Actual); Primary Completion 2023-02-20 (Actual); Study Completion 2023-02-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda Hanson, DC, MS, Study Director — University of Minnesota
Locations (2):
- United States (2):
  - University of Minnesota, Minneapolis, Minnesota
  - University of Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Supported Biopsychosocial Self-Management (SBSM) | Medical Care
Started | 20 | 22
Completed | 19 | 20
Not Completed | 1 | 2
Not completed — Lack of Efficacy | 1 | 0
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Supported Biopsychosocial Self-Management (SBSM) | Medical Care | Total
Number analyzed (Participants) | 20 | 22 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.3 (14.6) | 51.6 (14.0) | 52.9 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 14 | 25
  Male | 9 | 8 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 20 | 20 | 40
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 4 | 4
  White | 18 | 15 | 33
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Particpants Screened Per Month
Description: As a measure of recruitment feasibility, the average number of participants screened per month is reported
Time Frame: 6 month period of active study screening
Measure: Mean (Full Range); unit: participants per month
Groups:
- Screened Participants: Individuals contacting study staff expressing interest in participating
Arm/Group | Screened Participants
Number analyzed (Participants) | 617
participants per month | 103 [26 to 247]

2. Primary Outcome: Percentage of Screened Participants Who Are Female
Description: As a measure of recruitment feasibility, the number of female participants in the study is reported
Time Frame: 6 month period of active study screening
Measure: Count of Participants; unit: Participants
Arm/Group | Screened Participants
Number analyzed (Participants) | 617
Participants | 414

3. Primary Outcome: Percentage of Screened Participants Who Are From Racial or Ethnic Minority Populations
Description: As a measure of recruitment feasibility, the number of participants from racial or ethnic minority populations is reported.
Time Frame: 6 month period of active study screening
Measure: Count of Participants; unit: Participants
Arm/Group | Screened Participants
Number analyzed (Participants) | 617
Participants | 168

4. Primary Outcome: Number of Participants Enrolled Per Month
Description: As a measure of enrollment feasibility, the average number of participants recruited per month is reported.
Time Frame: 6 month period of active study screening
Measure: Mean (Full Range); unit: participants per month
Groups:
- Enrolled Participants: Individuals enrolled into the randomized trial
Arm/Group | Enrolled Participants
Number analyzed (Participants) | 42
participants per month | 7 [3 to 11]

5. Primary Outcome: Percentage of Enrolled Participants Who Are Female
Description: As a measure of enrollment feasibility, the number of female participants enrolled in the study is reported.
Time Frame: 6 month period of active study enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Enrolled Participants
Number analyzed (Participants) | 42
Participants | 25

6. Primary Outcome: Percentage of Enrolled Participants Who Are From Racial or Ethnic Minority Populations
Description: As a measure of enrollment feasibility, the number of participants enrolled from racial or ethnic minority populations is reported.
Time Frame: 6 month period of active enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Enrolled Participants
Number analyzed (Participants) | 42
Participants | 8

7. Primary Outcome: Percentage of Enrollees Not Receiving Any Treatment
Description: As a measure of intervention acceptability and credibility associated with feasibility, the number of enrollees not receiving any treatment is reported.
Time Frame: Through study treatment, an average of 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Supported Biopsychosocial Self-Management (SBSM) | Medical Care
Number analyzed (Participants) | 20 | 22
Participants | 0 | 1

8. Primary Outcome: Percentage of Enrollees Receiving Prohibited Treatments
Description: As a measure of intervention acceptability and credibility associated with feasibility, the number of enrollees receiving prohibited treatments, (contamination), during the 12-week intervention phase of the study is reported.
Time Frame: Through study treatment, an average of 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Supported Biopsychosocial Self-Management (SBSM) | Medical Care
Number analyzed (Participants) | 20 | 22
Participants | 1 | 1

9. Primary Outcome: Percentage of Enrollees Satisfied With Treatment
Description: As a measure of intervention acceptability and credibility associated with feasibility, treatment satisfaction was reported by participants via a 7-point Likert satisfaction scale, ranging from 1, "completely satisfied," to 7, "completely dissatisfied," where lower numbers indicate greater satisfaction. The percentage of enrollees satisfied with treatment is reported as a percent value representing those who choose "somewhat satisfied" or better on the scale.
Time Frame: Through study treatment, an average of 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Supported Biopsychosocial Self-Management (SBSM) | Medical Care
Number analyzed (Participants) | 20 | 22
Participants | 17 | 14

10. Primary Outcome: Percentage of Enrollees Attending Required Sessions
Description: As a measure of participant treatment adherence associated with feasibility, the number of enrollees attending the minimum number of required study sessions (6 for SBSM and 2 for Medical Care) are reported.
Time Frame: Through study treatment, an average of 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Supported Biopsychosocial Self-Management (SBSM) | Medical Care
Number analyzed (Participants) | 20 | 22
Participants | 19 | 20

11. Primary Outcome: Percentage of Enrollees in Supported Biopsychosocial Self-management Group Reporting Participation in Home Practice
Description: As a measure of participant treatment adherence associated with feasibility, the number of enrollees who are part of the supported biopsychosocial self-management arm of the study who self-report participation in home treatment practice is reported.
Time Frame: Through study treatment, an average of 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Supported Biopsychosocial Self-Management (SBSM)
Number analyzed (Participants) | 20
Participants | 19

12. Primary Outcome: Percentage of Enrollees in Medical Care Group Reporting Taking Medications as Prescribed
Description: As a measure of participant treatment adherence associated with feasibility, the number of enrollees who are part of the medical care arm self-reporting taking medications as prescribed is reported.
Time Frame: Through study treatment, an average of 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Medical Care
Number analyzed (Participants) | 22
Participants | 17

13. Primary Outcome: Percentage of Provider Visits Where All Required Intervention Activities Were Delivered
Description: As a measure of provider fidelity, the percentage of provider vists where 100% of required intervention activities were delivered is reported.
Time Frame: Through study treatment, an average of 3 months
Measure: Count of Units; unit: Visits
Units Other Than Participants: Visits
Arm/Group | Supported Biopsychosocial Self-Management (SBSM) | Medical Care
Number analyzed (Participants) | 20 | 22
Number analyzed (Visits) | 155 | 80
Visits | 111 | 79

14. Primary Outcome: Percentage of Enrollees Completing the Month 3 Assessment
Description: As a measure of data collection feasibility, the number of enrollees completing the month 3 assessment is reported.
Time Frame: Month 3 assessment
Measure: Count of Participants; unit: Participants
Arm/Group | Supported Biopsychosocial Self-Management (SBSM) | Medical Care
Number analyzed (Participants) | 20 | 22
Participants | 18 | 20

15. Primary Outcome: Percentage of Enrollees Completing the Month 6 Assessment
Description: As a measure of data collection feasibility, the number of enrollees completing the month 6 assessment is reported.
Time Frame: Month 6 assessment
Measure: Count of Participants; unit: Participants
Arm/Group | Supported Biopsychosocial Self-Management (SBSM) | Medical Care
Number analyzed (Participants) | 20 | 22
Participants | 18 | 20

16. Primary Outcome: Percentage of Weekly Pain Severity and Frequency Assessments Completed
Description: As a measure of data collection feasibility, the number of weekly pain severity and frequency assessments completed by participants is reported.
Time Frame: Through completion of all weekly assessments, an average of 6 months
Measure: Count of Units; unit: Weekly Surveys
Units Other Than Participants: Weekly Surveys
Arm/Group | Supported Biopsychosocial Self-Management (SBSM) | Medical Care
Number analyzed (Participants) | 20 | 22
Number analyzed (Weekly Surveys) | 520 | 572
Weekly Surveys | 461 | 479

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Supported Biopsychosocial Self-Management (SBSM) | Medical Care
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/20 | 2/22
Other Adverse Events (participants affected / at risk) | 12/20 | 14/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Supported Biopsychosocial Self-Management (SBSM) (N=20) | Medical Care (N=22)
Fracture injury after fall (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Supported Biopsychosocial Self-Management (SBSM) (N=20) | Medical Care (N=22)
Back problems - soreness/stiffness (Musculoskeletal and connective tissue disorders) | 7 (10) | 5 (8)
Back problems - new back or leg pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 6 (8)
Back problems - increased back or leg pain (Musculoskeletal and connective tissue disorders) | 5 (6) | 8 (11)
Back problems - numbness or tingling (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Gastrointestinal problems - dry mouth (Gastrointestinal disorders) | 1 (1) | 3 (3)
Gastrointestinal problems - indigestion (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastrointestinal problems - abdominal pain (Gastrointestinal disorders) | 2 (2) | 4 (4)
Gastrointestinal problems - reflux (Gastrointestinal disorders) | 0 (0) | 3 (3)
Gastrointestinal problems - constipation (Gastrointestinal disorders) | 3 (5) | 2 (2)
Gastrointestinal problems - decreased appetite (Gastrointestinal disorders) | 0 (0) | 2 (2)
Mental health problems - emotional discomfort (General disorders) | 3 (4) | 1 (1)
Other problems - headache (Nervous system disorders) | 2 (2) | 3 (5)
Other problems - breathing problems (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Other problems - rash (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Other problems - blurry vision or vision loss (Eye disorders) | 0 (0) | 2 (4)
Other problems - sleep problems (General disorders) | 3 (3) | 5 (6)
Other problems - drowsiness (General disorders) | 3 (3) | 4 (5)
Other problems - weight gain or loss (General disorders) | 2 (2) | 4 (6)
Other problems - bowel or bladder changes (General disorders) | 2 (3) | 3 (3)
Other problems - bruising (General disorders) | 0 (0) | 3 (3)
Other problems - weakness (General disorders) | 2 (2) | 2 (4)
Other problems - clumsiness (General disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-07-18): https://cdn.clinicaltrials.gov/large-docs/21/NCT05022121/Prot_SAP_001.pdf
  • Informed Consent Form (2021-07-19): https://cdn.clinicaltrials.gov/large-docs/21/NCT05022121/ICF_000.pdf